CLINICAL TRIAL: NCT00294307
Title: Hospital to Home: Cognitively Impaired Elders/Caregivers
Brief Title: Enhancing Care Coordination: Hospital to Home for Cognitively Impaired Older Adults and Their Caregivers
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Other Study IDs: R01AG023116 (NIH); R01AG023116 (NIH)
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Dementia; Dementia, Vascular; Alzheimer Disease; Delirium, Dementia, Amnestic, Cognitive Disorders; Lewy Body Disease; Mild Cognitive Impairment
Keywords: Nursing Models of Care; Collaborative Care; Care Management; Transitional Care; Advanced Practice Nurse Care Interventions; Cognitive Impairment; Dementia; Delirium
MeSH Terms: conditions — Dementia; Dementia, Vascular; Alzheimer Disease; Neurocognitive Disorders; Lewy Body Disease; Cognitive Dysfunction; Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Advanced Practice Nurse Care (APNC): Hospital to Home
  Interventions: Behavioral: Advanced Practice Nurse Care (APNC)
- Augmented Standard Care (ASC): Hospital only
  Interventions: Behavioral: Augmented Standard Care (ASC)
- Resource Nurse Care (RNC): Hospital only
  Interventions: Behavioral: Resource Nurse Care (RNC)

INTERVENTIONS:
Behavioral: Augmented Standard Care (ASC) — Standard hospital care and, if referred, home care plus early identification of CI during the patients' hospitalization by trained research assistants with immediate verbal feedback and documentation to patients' primary nurses, attending physicians and discharge planners [low intensity];
  Groups: Augmented Standard Care (ASC)
Behavioral: Resource Nurse Care (RNC) — Standard hospital and, if referred, home care plus early identification of CI during the patient's hospitalization (ASC) and hospital care by RNs trained in the use of expert clinical guidelines developed to enhance the care management of hospitalized cognitively impaired elders and to facilitate their transition from hospital to home [medium intensity];.
  Groups: Resource Nurse Care (RNC)
Behavioral: Advanced Practice Nurse Care (APNC) — Standard hospital care plus ASC and transitional care starting in the hospital and substituting for standard home care and provided by Advanced Practice Nurses (APNs) with advanced training in the management of CI patients using an evidence-based protocol designed specifically for this patient group and their caregivers [high intensity].
  Groups: Advanced Practice Nurse Care (APNC)

SUMMARY:
Aim 1. To compare across three hospital sites the effects on health and cost outcomes observed by the following three interventions, each designed to enhance adaptation and improve outcomes of hospitalized cognitively impaired elders and their caregivers:

1. augmented standard care (ASC) - standard hospital and, if referred, home care plus early identification of CI during the patients' hospitalization by trained registered nurses (RNs) with immediate feedback to patients' primary nurses, attending physicians and discharge planners;
2. resource nurse care (RNC) - standard hospital and, if referred, home care plus early identification of CI during the patient's hospitalization by trained RNs and hospital care by RNs trained in the use of expert clinical guidelines developed to enhance the care management of hospitalized cognitively impaired elders and to facilitate their transition from hospital to home; or,
3. advanced practice nurse care (APNC) - standard hospital care plus transitional (hospital to home) care substituting for standard home care and provided by APNs with advanced training in the management of CI patients using an evidence-based protocol designed specifically for this patient group and their caregivers.

[H1] We hypothesize that health and cost outcomes with APNC, a comprehensive intervention designed to meet the unique needs of cognitively impaired older adults hospitalized for an acute medical or surgical event and their caregivers will be associated, relative to health and cost outcomes with ASC and RNC, with improvement in patient, caregiver and cost outcomes.

[H2] We hypothesize that improvements in patient, caregiver and cost outcomes observed for the RNC group will be greater than those observed for the ASC group.

Aim 2. To compare within each site and over time, health and cost outcomes (identified in Aim 1) from patients treated with either ASC or RNC, both relatively lower intensity interventions, with the outcomes of patients at the same site observed after switching to APNC, a high intensity intervention.

[H3] We hypothesize that compared to patients receiving the ASC or the RNC interventions, patients at the same site will have improved patient, caregiver and cost outcomes after the site switches to APNC.

[H4] We hypothesize that patient, caregiver and cost outcomes achieved by the groups receiving APNC interventions at T1 and T2 will be similar.

DETAILED DESCRIPTION:
Cognitive impairment (CI) is a major health problem complicating the care of increasing numbers of older adults hospitalized for an acute medical or surgical condition. Dementia and delirium, the most common causes of CI among these elders, is associated with higher mortality rates, increased morbidity and higher health care costs. A growing body of science suggests that these patients and their caregivers are particularly vulnerable to systems of care that either do not recognize or ignore their needs. The consequences are devastating for the patients and their caregivers and add tremendous burden to hospital staffs coping with a severe shortage of nurses. For these reasons, the Institute of Medicine identified improved care management of this patient group as a national priority for action. Unfortunately, little evidence is available to guide optimal care of this patient group or to address the unique needs of their caregivers. Collectively, available evidence suggests that these patients may benefit from interventions aimed at improving management of CI, comorbid conditions or both but the exact nature and intensity of intervention needed to effectively and efficiently improve their outcomes and those of their caregivers is not known. Thus, the timing is excellent for rigorous research aimed at identifying care management strategies that will result in high quality, cost-effective outcomes for this challenging patient group and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 65 and older
* Speaks English
* Resides within 30 miles of admitting hospital site
* Admitted from home to one of three hospital sites
* a documented history of pre-existing dementia in their medical records or pre-screen positive for cognitive impairment using our Pre-Screen Process.
* a primary caregiver (knowledgeable informant), defined as the spouse, family member, partner or friend, who will provide support following discharge to home and is reachable by telephone.

Exclusion Criteria:

* End Stage Disease
* Active untreated substance abuse or psychiatric conditions
* Primary cancer diagnosis (active treatment)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Hospitalized community dwelling older adults with cognitive impairment and a caregiver
Sampling Method: Non-Probability Sample
Enrollment: 814 (Actual)
Dates: Start 2006-02; Primary Completion 2010-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Patient - Function | At hospital admission and at 2-, 6-, 12-, and 26-weeks post-discharge
  Basic Activities of Daily Living
Caregiver - Burden | At hospital admission and at 2-, 6-, 12-, and 26-weeks post-discharge
Patient - Health Care Costs | Through 6 months
Patient - Time to first rehospitalization or death; total rehospitalization days | From index hospital discharge through 6 months
  Time calculated from index hospital discharge to first rehospitalization or death. Total days rehospitalized through six months.

SECONDARY OUTCOMES:
Patient - Total rehospitalizations | From index hospital discharge through 6 months
Patient - Cognitive Function | At hospital admission and at 2-, 6-, 12-, and 26-weeks post-discharge
Patient - Care Management | From enrollment through 6 months
Patient - Symptoms (Physical and depressive symptoms) | At hospital admission and at 2-, 6-, 12-, and 26-weeks post-discharge
Patient - Neuropsychiatric Behaviors | At hospital admission and at 2-, 6-, 12-, and 26-weeks post-discharge
Patient - Quality of Life | At hospital admission and at 2-, 6-, 12-, and 26-weeks post-discharge
Patient/Caregiver - Satisfaction with care | At 2-weeks and post APNC intervention
Caregiver - Depressive Symptoms | At hospital admission and at 2-, 6-, 12-, and 26-weeks post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Mary D Naylor, PhD, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn-Presbyterian Medical Center, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Naylor MD, Hirschman KB, Bowles KH, Bixby MB, Konick-McMahan J, Stephens C. Care coordination for cognitively impaired older adults and their caregivers. Home Health Care Serv Q. 2007;26(4):57-78. doi: 10.1300/j027v26n04_05. PMID 18032200
- [Background] Naylor MD, Stephens C, Bowles KH, Bixby MB. Cognitively impaired older adults: from hospital to home. Am J Nurs. 2005 Feb;105(2):52-61; quiz 61-2. doi: 10.1097/00000446-200502000-00028. No abstract available. PMID 15674058
- [Background] McCauley K, Bradway C, Hirschman KB, Naylor MD. Studying nursing interventions in acutely ill, cognitively impaired older adults. Am J Nurs. 2014 Oct;114(10):44-52. doi: 10.1097/01.NAJ.0000454851.22018.5d. PMID 25251126
- [Background] Shankar KN, Hirschman KB, Hanlon AL, Naylor MD. Burden in caregivers of cognitively impaired elderly adults at time of hospitalization: a cross-sectional analysis. J Am Geriatr Soc. 2014 Feb;62(2):276-84. doi: 10.1111/jgs.12657. Epub 2014 Feb 6. PMID 24502827
- [Background] Hirschman KB, Paik HH, Pines JM, McCusker CM, Naylor MD, Hollander JE. Cognitive Impairment among Older Adults in the Emergency Department. West J Emerg Med. 2011 Feb;12(1):56-62. PMID 21691473
- [Result] Bradway C, Trotta R, Bixby MB, McPartland E, Wollman MC, Kapustka H, McCauley K, Naylor MD. A qualitative analysis of an advanced practice nurse-directed transitional care model intervention. Gerontologist. 2012 Jun;52(3):394-407. doi: 10.1093/geront/gnr078. Epub 2011 Sep 9. PMID 21908805
- [Result] Naylor MD, Hirschman KB, Hanlon AL, Bowles KH, Bradway C, McCauley KM, Pauly MV. Comparison of evidence-based interventions on outcomes of hospitalized, cognitively impaired older adults. J Comp Eff Res. 2014 May;3(3):245-57. doi: 10.2217/cer.14.14. PMID 24969152
- [Result] Naylor MD, Hirschman KB, Hanlon AL, Bowles KH, Bradway C, McCauley KM, Pauly MV. Effects of alternative interventions among hospitalized, cognitively impaired older adults. J Comp Eff Res. 2016 May;5(3):259-72. doi: 10.2217/cer-2015-0009. Epub 2016 May 5. PMID 27146416
- [Result] Pauly MV, Hirschman KB, Hanlon AL, Huang L, Bowles KH, Bradway C, McCauley K, Naylor MD. Cost impact of the transitional care model for hospitalized cognitively impaired older adults. J Comp Eff Res. 2018 Sep;7(9):913-922. doi: 10.2217/cer-2018-0040. Epub 2018 Sep 11. PMID 30203668